CLINICAL TRIAL: NCT01942044
Title: Impact of Stent Platform on Shear Stress Distribution and Subsequent Vessel Healing After Drug-eluting Stent Implantation (SHEAR DES)
Brief Title: Relation Among Shear Stress Distribution, Stent Design, and Subsequent Vessel Healing After Drug-eluting Stent Implantation (SHEAR DES)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Hiromasa Otake, Assistant Professor, Kobe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOtake1
Record Dates: First submitted 2013-09-07; First posted 2013-09-13 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Heart Disease
Keywords: Shear stress; Optical coherence tomography; Drug-eluting stents
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Promus element (Experimental): Promus element is a thin struts, 2-link design, evelolimus-eluting stents.
  Interventions: Device: Promus element, Xience prime, and Nobori
- Xience Prime (Active Comparator): Xience Prime is a thin struts, 3-link design, evelolimus-eluting stents.
  Interventions: Device: Promus element, Xience prime, and Nobori
- Nobori (Active Comparator): Nobori is a thick struts, 2-link design, biolimus-eluting stents.
  Interventions: Device: Promus element, Xience prime, and Nobori

INTERVENTIONS:
Device: Promus element, Xience prime, and Nobori

SUMMARY:
The purpose of this study is to evaluate the differences of wall shear stress distribution among different types of drug-eluting stents and its impact on vessel healing evaluated by intravascular optical coherence tomography evaluation.

DETAILED DESCRIPTION:
Background: Distribution of wall shear stress (WSS) may be different according to stent designs. The impact of WSS after stent implantation may impact future vessel healing after current generation drug-eluting stents implantation. Although previous studies used IVUS (intravascular ultrasound) and angiography to determine WSS from computational fluid dynamics (CFD) simulations, new methods using higher resolution OCT (optical coherence tomography) are warranted to further evaluate the impact of stent design on WSS with current generation drug-eluting stents.

Methods: For these purpose, we will enroll a total of 30 patients with stable angina who are scheduled for percutaneous coronary intervention. Those patients were randomized to thin-strut (81μm) 2-link Promus element (PE: n=10), thin-strut (81μm) 3-link Xience Prime (XP: n=10), or thick-strut (145μm) 2-link Nobori stents (NO: n=10) and underwent OCT and coronary CT angiography (CTA) after stenting. Post stent WSS was calculated using CFD simulations based on patient-specific reconstructed 3D arteries created by the fusion of OCT and CTA data, normalized using WSS in the proximal unstented region. Also, follow-up angiography and OCT are performed for the assessment of vessel healing as well as WSS distribution 8months after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old.
* Indication of PCI with Xience prime, Nobori, or Promus element.
* Clinical diagnosis of stable angina, unstable angina or silent ischemia with reference vessel diameters ranging from 2.5-3.5mm.
* Underwent CT angiography before PCI.
* To agree to review and record all the clinical course in this research protocol.

Exclusion Criteria:

* Previous history of pancytopenia, liver function, renal dysfunction, hypersensitive history of the drug.
* Low ejection fraction (LVEF<=30%), an impaired liver function, and renal dysfunction (eGFR<=40)
* Severe calcification
* Stent restenosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of uncovered struts | 8 months

SECONDARY OUTCOMES:
Neointimal thickness | 8 months
The percentage of malapposed struts | 8 months
Area of low wall shear stress | Baseline
  Baseline area of low wall shear stress will be calculated within 1 month after obtaining post stent OCT and CTA images.
Area of high oscillatory shear index | Baseline
  Baseline area of high oscillatory shear index will be calculated within 1 month after obtaining post stent OCT and CTA images.
Area of low wall shear stress | 8 months
Area of high oscillatory shear index | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Hiromasa Otake, MD, PhD, Principal Investigator — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Kobe, Hyōgo, Japan